CLINICAL TRIAL: NCT04730453
Title: Electromagnetic Navigation Bronchoscopy Guided Ablation Therapy Combined With VATS in the Treatment of Multiple Primary Lung Cancers
Brief Title: ENB-guided Ablation Therapy Combined With VATS in the Treatment of MPLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Other Study IDs: SHCHE202101
Record Dates: First submitted 2021-01-24; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer
Keywords: Electromagnetic Navigation Bronchoscopy (ENB); Video-Assisted Thoracic Surgery (VATS); Multiple Primary Lung Cancers (MPLC); Ablation Therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ENB-guided ablation therapy combined with VATS — After receiving multidisciplinary assessments, Lesion A will receive ENB-guided ablation therapy and Lesion B will receive VATS at the same time.

SUMMARY:
The study is designed as a prospective trial whose purpose is to evaluate the effectiveness and safety of ENB-guided ablation therapy combined with VATS in the treatment of multiple primary lung cancers (MPLC).

DETAILED DESCRIPTION:
Patients will be first screened, and only after meeting all the selection criteria, not meeting any exclusion criteria, and signing the informed consent, could they be enrolled in the group to receive ENB-guided ablation therapy combined with VATS. The primary endpoint is objective response rate (ORR). The secondary endpoints include progression-free survival (PFS), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. The subject is diagnosed as multiple primary lung cancer via preoperative imaging/pathological examination.
3. Thin-slice CT images show that the ablation Lesion A is accessible/adjacent to bronchi and the size is ≤ 3 cm.
4. The subject with multiple primary lung cancers can be treated with ENB-guided ablation therapy combined with VATS according to multidisciplinary assessment.

Exclusion Criteria:

1. The subject who cannot tolerate general anesthesia for their cardiopulmonary function, or there are other contraindications, such as uncorrectable coagulopathy.
2. The situation in which the investigators think that the subject is not suitable to participate in this study.

Min Age: 18 Minutes | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet inclusion/exclusion will be enrolled in the study consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of ablation efficacy, ORR (objective response rate) | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 years.
  ORR is defined as the proportion of patients with complete response (CR) and partial response (PR) after ablation therapy. Efficacy evaluation is based on Modifield Response Evaluation Criteria in Solid Tumors (mRECIST).

SECONDARY OUTCOMES:
Evaluation of ablation efficacy, PFS (progression-free survival) | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  PFS is defined as the time from the start of treatment to the first occurrence of disease progression or death for any cause.
Evaluation of ablation efficacy, OS (overall survival) | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  OS is defined as the time from the start of treatment to the death of the patient.
Observation of complications of ablation | From date of treatment to the one month after ablation.
  Complications refer to the combination of serious adverse events related to the operation during or after the operation, mainly including pneumothorax and bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howington JA, Blum MG, Chang AC, Balekian AA, Murthy SC. Treatment of stage I and II non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e278S-e313S. doi: 10.1378/chest.12-2359. PMID 23649443
- [Background] Ambrogi MC, Fanucchi O, Dini P, Melfi F, Davini F, Lucchi M, Massimetti G, Mussi A. Wedge resection and radiofrequency ablation for stage I nonsmall cell lung cancer. Eur Respir J. 2015 Apr;45(4):1089-97. doi: 10.1183/09031936.00188014. Epub 2015 Feb 19. PMID 25700387
- [Background] Ye X, Fan W, Wang H, Wang J, Wang Z, Gu S, Feng W, Zhuang Y, Liu B, Li X, Li Y, Li C, Xiao Y, Yang P, Yang X, Yang W, Chen J, Zhang R, Lin Z, Meng Z, Hu K, Liu C, Peng Z, Han Y, Jin Y, Lei G, Zhai B, Huang G. Expert consensus workshop report: Guidelines for thermal ablation of primary and metastatic lung tumors (2018 edition). J Cancer Res Ther. 2018;14(4):730-744. doi: 10.4103/jcrt.JCRT_221_18. PMID 29970646
- [Background] Harris K, Puchalski J, Sterman D. Recent Advances in Bronchoscopic Treatment of Peripheral Lung Cancers. Chest. 2017 Mar;151(3):674-685. doi: 10.1016/j.chest.2016.05.025. Epub 2016 Jun 10. PMID 27292045
- [Background] Tsushima K, Koizumi T, Tanabe T, Nakagawa R, Yoshikawa S, Yasuo M, Kubo K. Bronchoscopy-guided radiofrequency ablation as a potential novel therapeutic tool. Eur Respir J. 2007 Jun;29(6):1193-200. doi: 10.1183/09031936.00111306. Epub 2007 Mar 14. PMID 17360727
- [Background] Tanabe T, Koizumi T, Tsushima K, Ito M, Kanda S, Kobayashi T, Yasuo M, Yamazaki Y, Kubo K, Honda T, Kondo R, Yoshida K. Comparative study of three different catheters for CT imaging-bronchoscopy-guided radiofrequency ablation as a potential and novel interventional therapy for lung cancer. Chest. 2010 Apr;137(4):890-7. doi: 10.1378/chest.09-1065. Epub 2009 Oct 26. PMID 19858232
- [Background] Xie F, Zheng X, Xiao B, Han B, Herth FJF, Sun J. Navigation Bronchoscopy-Guided Radiofrequency Ablation for Nonsurgical Peripheral Pulmonary Tumors. Respiration. 2017;94(3):293-298. doi: 10.1159/000477764. Epub 2017 Jul 6. PMID 28683443